CLINICAL TRIAL: NCT02484651
Title: Can Adequacy of Anesthesia Depth and Quality of Recovery be Influenced by the Level of Neuromuscular Blockade: a Randomized Controlled Study Assessing Propofol and Remifentanil Requirements and Quality of Recovery in Patients With a Standard Practice of Non-deep Rocuronium Neuromuscular Blockade Versus Deep Neuromuscular Blockade Reversed With Sugammadex
Brief Title: Can Adequacy of Anesthesia Depth and Quality of Recovery be Influenced by the Level of Neuromuscular Blockade?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Hospitalar do Porto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Pedro Amorim, MD, Pedro Amorim, MD, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014.145; 2014-005238-76 (EudraCT Number)
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Neuromuscular Block
Keywords: deep neuromuscular block; sugammadex; stability of anesthesia; suppression of EMG activity; PQRS; General Anesthesia; Quality of Recovery
MeSH Terms: interventions — Sugammadex; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Group (No Intervention): Standard Clinical Practice Group - standard neuromuscular block, with a standard rocuronium dose for intubation (0.6 mg/kg). If required, the reversal of neuromuscular block is performed with neostigmine.
- Deep NMB group (Experimental): Deep Neuromuscular Block group - with a standard rocuronium dose for intubation (0.6 mg/kg), followed by a constant infusion of rocuronium (10-15 ug/kg/min) to guarantee a PTC less or equal to 2 on the TOF monitor (PTC is evaluated every 5 minutes). The reversal of neuromuscular block is performed with Sugammadex (4 mg/kg).
  Interventions: Drug: Sugammadex; Drug: Rocuronium

INTERVENTIONS:
Drug: Sugammadex — Reversal of deep neuromuscular block
  Other Names: Org 25969; Bridion
  Arms: Deep NMB group
Drug: Rocuronium — Maintenance of deep neuromuscular block
  Other Names: Zemuron; Esmeron
  Arms: Deep NMB group

SUMMARY:
The investigators hypothesize that an anesthetic protocol maintaining deep neuromuscular block throughout the entire surgical procedure followed by sugammadex reversal, would suppress EMG activity and result in improved anesthetic stability by reducing the variability of the Bispectral Index of the EEG, and be beneficial by reducing the total doses of the anesthetic drugs propofol and remifentanil required to maintain an adequate level of anesthesia (BIS between 40 and 60).

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I-III
* Between 18 - 80 years old
* Scheduled for routine cervical surgery
* Minimum duration of surgery is 90 minutes and performed with total intravenous anaesthesia (TIVA) with the hypnotic propofol, the analgesic remifentanil and the neuromuscular relaxant rocuronium
* Patients that are able to and do provide a signed informed consent form

Exclusion Criteria:

* Patients with neuromuscular diseases and severe cardiac and respiratory pathologies
* Contra indication for any of the drugs used
* Not able to complete the baseline PQRS test.
* Indication to perform tracheal intubation using fibroscopy
* Patients who are pregnant or nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06-28 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Amorim, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar do Porto, Porto, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on the 2016/9/19 and finished on 2017/6/28 at Centro Hospitalar do Porto, Portugal.
Pre-assignment Details: 3 patients were excluded from the study after screening (signing the informed consent) but before randomization and assignment to the groups, due to:
  * 2 patients had their surgery postponed less than 2 hours before the schedule time
  * the scheduled surgical position of 1 patient was altered by the surgeon just before the start of the procedure.
Period: Overall Study
Arm/Group | Standard Group | Deep NMB Group
Started | 35 (35 patients were randomized) | 35 (35 patients were randomized)
End of Clinical Study (Patients that followed the protocol and finished the clinical study.) | 35 | 35
Data Analysis (Patients with valid recorded data included in the data analysis) | 32 | 31
Completed | 32 | 31
Not Completed | 3 | 4
Not completed — Patients' data files were corrupted. | 1 | 1
Not completed — BIS monitoring failed. | 1 | 1
Not completed — Time of the procedure less than 90 min. | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Group | Deep NMB Group | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.7) | 52.6 (7.9) | 52.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 31 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Portugal | 32 | 31 | 63
Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] | 105.6 (12.8) | 101.4 (12.5) | 103.5 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: BIS Signal Variability Using the Measured Standard Deviation During the Maintenance Phase of Anesthesia
Description: BIS (Bispetral Index of the EEG) sample standard deviation during the maintenance phase of anesthesia was used as a measure of signal variability, maintenance phase is defined as the time between the first time the BIS signal drops below 60 after loss of consciousness, until the time the BIS signal goes above 60 after the propofol infusion is stopped. BIS signal varies between 0 to 100. BIS values near 100 represent an "awake" clinical state while 0 denotes the maximal effect an isoelectric EEG. The aim was to maintain the BIS value within a target range of 40 to 60. The higher the BIS sample standard deviation the higher the oscillation around the sample mean.
Time Frame: Maintenance of anesthesia, an average of 130 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Group | Deep NMB Group
Number analyzed (Participants) | 32 | 31
units on a scale | 7.6 (1.6) | 7.8 (1.6)
Statistical Analysis 1: Comparison: Standard Group vs Deep NMB Group; Sample size calculation was performed with a power of 0.80 and an α of 0.05, considering the primary hypothesis of a reduction in the BIS variability (measured as the standard deviation). A 25% reduction on the BIS variability (standard deviation) was considered clinically relevant, and gave a minimum sample size of 26 per group; Test type: Superiority; p = 0.651, t-test, 2 sided

2. Primary Outcome: Required Effect-site Concentrations of Propofol and Remifentanil
Description: Mean effect-site concentration of propofol required during maintenance of anesthesia (using target controlled infusion).
  Mean effect-site concentration of remifentanil required during maintenance of anesthesia (using target controlled infusion).
Time Frame: Maintenance of anesthesia, an average of 130 minutes
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Deep NMB Group: Deep Neuromuscular Block group - with a standard rocuronium dose for intubation (0.6 mg/kg), followed by a constant infusion of rocuronium (10-15 ug/kg/min) to guarantee a PTC(Post-Tetanic-Count) less or equal to 2 on the TOF(Train of Four) monitor (PTC is evaluated every 5 minutes). The reversal of neuromuscular block is performed with Sugammadex (4 mg/kg).
  Sugammadex: Reversal of deep neuromuscular block
  Rocuronium: Maintenance of deep neuromuscular block
Arm/Group | Standard Group | Deep NMB Group
Number analyzed (Participants) | 32 | 31
ng/ml
  Propofol | 3000 (560) | 2450 (550)
  Remifentanil | 3.26 (1.02) | 2.84 (1.12)
Statistical Analysis 1: Comparison: Standard Group vs Deep NMB Group; This statistical analysis applies to the propofol effect-site concentration. Sample size calculation was performed with a power of 0.80 and an α of 0.05 also a reduction in the propofol drug consumption (measured as the average effect-site concentration) during maintenance of anesthesia. A reduction on propofol mean effect-site concentration of 20% was considered clinically relevant, giving a minimum of 34 patients per group; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Standard Group vs Deep NMB Group; This statistical analysis applies to the remifentanil effect-site concentration. Sample size calculation was performed with a power of 0.80 and an α of 0.05 also a reduction in the remifentanil drug consumption (measured as the average effect-site concentration) during maintenance of anesthesia. A reduction on on remifentanil average effect-site concentration of 20% was considered clinically relevant, giving a minimum of 24 patients per group; Test type: Superiority; p = 0.245, t-test, 2 sided

3. Secondary Outcome: PQRS Results at 15 and 40 Minutes After Surgery (Taking Into Account the Patient Baseline Values of the PQRS Test Done on the Preanesthetic Visit)
Description: PQRS(Post-operative Quality Recovery Scale) recovery rate at 15 minutes post surgery and PQRS recovery rate at 40 minutes post surgery. Recovery is defined as returning to PQRS baseline values.
Time Frame: 15 and 40 minutes after surgery
Population: 10 patients were not able to complete the PQRS test at 15 minutes, since they were not able to communicate or understand the questions.
  1 patient was not able to complete the PQRS test at 15 and 40 minutes due to problems in the vocal cords.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Group | Deep NMB Group
Number analyzed (Participants) | 32 | 31
Participants
  15 minutes: number analyzed (Participants) | 26 | 26
  15 minutes: Overall recovery | 2 | 5
  15 minutes: Did not recovered | 24 | 21
  40 minutes: number analyzed (Participants) | 32 | 30
  40 minutes: Overall recovery | 0 | 3
  40 minutes: Did not recovered | 32 | 27
Statistical Analysis 1: Comparison: Standard Group vs Deep NMB Group; The null hypothesis was that PQRS overall recovery at 15 minutes was independent from the study group; Test type: Superiority; p = 0.419, Fisher Exact
Statistical Analysis 2: Comparison: Standard Group vs Deep NMB Group; The null hypothesis was that PQRS overall recovery at 40 minutes was independent from the study group; Test type: Superiority; p = 0.107, Fisher Exact

4. Secondary Outcome: PQRS Satisfaction Results at Day 3 After Surgery
Description: Patient satisfaction with anesthetic care rated as: Not satisfied, A little satisfied, Moderately satisfied ,Satisfied, Totally Satisfied
Time Frame: 3rd day after surgery
Population: 4 patients did not complete the questionnaire on the 3rd day, since they did not pick up the phone.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Group | Deep NMB Group
Number analyzed (Participants) | 30 | 29
Participants
  Totally satisfied | 27 | 27
  Satisfied | 3 | 2
  Moderately satisfied | 0 | 0
  A little satisfied | 0 | 0
  Not satisfied | 0 | 0
Statistical Analysis 1: Comparison: Standard Group vs Deep NMB Group; The null hypothesis was that PQRS satisfaction with anesthetic care was independent of the study group; Test type: Superiority; p = 0.669, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were collected by the researchers up to 3 days after surgery.
Arm/Group | Standard Group | Deep NMB Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 6/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Group (N=35) | Deep NMB Group (N=35)
Emergence delirium (Nervous system disorders) | 0 (0) | 2 (2)
Neck pain (Surgical and medical procedures) | 1 (1) | 0 (0) — Neck pain after discharge
Nausea and urinary retention (General disorders) | 1 (1) | 0 (0) — Nausea and urinary retention in the recovery
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Tachycardia of 120bpm in the recovery
Post-operative hypertension (General disorders) | 0 (0) | 1 (1) — Post-operative hypertension in the recovery room (Systolic Pressure 220 mmHg)
Asystole of 20 seconds (Cardiac disorders) | 0 (0) | 1 (1) — Asystole of 20 seconds during laryngoscopy resolved with IV atropine
Post-operative dyspnea and anxiety (Surgical and medical procedures) | 0 (0) | 1 (1) — Post-operative dyspnea and anxiety, shown on ENT examination, to have been caused by vocal cord paralysis due to a surgical complication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT02484651/Prot_SAP_000.pdf